CLINICAL TRIAL: NCT04259515
Title: Randomized Multicentric Trial to Compare Efficacy and Security of Bucberg vs Del Nido Cardioplegic Solutions in Isolated Aortic Valve Replacement.
Brief Title: Buckberg vs Del Nido in Isolated Aortic Valve Replacement
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IIBSP-CAR-2018-71; 2018-002701-59 (EudraCT Number)
Record Dates: First submitted 2020-01-21; First posted 2020-02-06 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Cardiac Surgical Procedures
MeSH Terms: interventions — Del Nido cardioplegia solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bukcberg (Active Comparator): Buckberg cardioplegical solution administered antegrade and/or retrograde at 1-2ml/Kg for cardiac arrest induction. Arrest manteinance with antegrade and/or retrograde administration at 1-2ml/Kg every 15 to 20 minutes. Reperfusion dose with antegrade or retrograde administration at 15-20 ml/Kg before removing the aortic crossclamp.
  Interventions: Drug: Buckberg
- Del Nido (Experimental): Del Nido cardioplegic solution administered in a single dose at 15-20mg/Kg with a maximum dose of 1L of solution, administered antegrade or retrograde. In those patients in wich the crossclamping time exceed 90 to 120 minutes a manteinance dose of 500ml will be administered.
  Interventions: Drug: Del Nido

INTERVENTIONS:
Drug: Del Nido — Del Nido cardioplegic solution administered in a single dose at 15-20mg/Kg with a maximum dose of 1L of solution, administered antegrade or retrograde. In those patients in wich the crossclamping time exceed 90 to 120 minutes a manteinance dose of 500ml will be administered.
  Arms: Del Nido
Drug: Buckberg — Buckberg cardioplegical solution administered antegrade and/or retrograde at 1-2ml/Kg for cardiac arrest induction. Arrest manteinance with antegrade and/or retrograde administration at 1-2ml/Kg every 15 to 20 minutes. Reperfusion dose with antegrade or retrograde administration at 15-20 ml/Kg before removing the aortic crossclamp.
  Arms: Bukcberg

SUMMARY:
The study compares safety and efficacy of the Del Nido cardioplegic solution, comparing it with the Buckberg cardioplegic solution in single aortic valve replacement procedures. Half the patients will receive the Del Nido solutions while the other half will receive the Buckberg solution.

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years old
* Patients listed for elective aortic valve replacement
* Patients that have signed informed consent

Exclusion Criteria:

* Emergent surgery
* Patients that do not accept blood transfusion
* Patients with previous cardiac surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 286 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Mortality | 30 days
  All cause mortality
Troponin T | 5 days
  Troponin T blood levels
CK | 5 days
  CK blood levels

CONTACTS AND LOCATIONS:
Overall Officials: Manel Tauron, MD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (2):
- Spain (2):
  - Hospital Germans Trias i Pujol, Badalona, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona

IPD SHARING:
Plan to Share IPD: Yes